CLINICAL TRIAL: NCT04638985
Title: A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Immunogenicity and Safety of Combined Immunization of Sabin-strain Inactivated Polio Vaccine (sIPV), Diphtheria, Tetanus, Pertussis Vaccine (DTaP) and Measles, Moms and Rubella Vaccine (MMR)
Brief Title: Evaluation of Immunogenicity and Safety of Combined Immunization of sIPV, DTaP and MMR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network); Anhui Provincial Center for Disease Control and Prevention (Unknown); Sichuan Center for Disease Control and Prevention (Other Government); Beijing Institute of Biological Products Co Ltd. (Industry); Chengdu Institute of Biological Products Co.,Ltd. (Industry); Peking University (Other); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sIPV-DTaP-MMR-2020
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (sIPV+DTaP+MMR) (Experimental): 150 subjects; simultaneously administration of sIPV+DTaP+MMR as booster immunization at the age of 18 months old, 0.5 ml each, respectively
  Interventions: Biological: sIPV+DTaP+MMR
- group 2 (sIPV) (Active Comparator): 150 subjects; vaccination of 0.5 ml sIPV as booster immunization at the age of 18 months old
  Interventions: Biological: sIPV
- group 3 (DTaP) (Active Comparator): 150 subjects; vaccination of 0.5 ml DTaP as booster immunization at the age of 18 months old
  Interventions: Biological: DTaP
- group 4 (MMR) (Active Comparator): 150 subjects; vaccination of 0.5 ml MMR as booster immunization at the age of 18 months old
  Interventions: Biological: MMR

INTERVENTIONS:
Biological: sIPV+DTaP+MMR — sIPV+DTaP+MMR at the age of 18 month old
  Arms: group 1 (sIPV+DTaP+MMR)
Biological: sIPV — sIPV at the age of 18 month old
  Arms: group 2 (sIPV)
Biological: DTaP — DTaP at the age of 18 month old
  Arms: group 3 (DTaP)
Biological: MMR — MMR at the age of 18 month old
  Arms: group 4 (MMR)

SUMMARY:
Eligible,healthy infants who have finished the 3-dose-schedule of sIPV+DTaP combined vaccination clinical trial (NCT04054882) will be recruited and divided into 4 groups, and will receive vaccination at the age of 18-month-old as follows:

Group 1: sIPV + DTaP + MMR, Group 2: sIPV only, Group 3: DTaP only, Group 4: MMR only.

The immunogenicity and safety of the 4 groups will be compared and analyzed before and 30 days after vaccination.

DETAILED DESCRIPTION:
Following the clinical trial of "Combined Immunization of sIPV and DTaP" in 2019, this study recruits 600 18-month-old subjects who have received 3 doses of sIPV + DTaP, and gives them a 4th dose of vaccination (booster immunization). They are divided into 4 different groups, with 150 subjects in each group, and are innoculated with different vaccines.

To be specific, group 1 receives sIPV (0.5ml)+ DTaP (0.5ml)+ MMR(0.5ml); group 2 receives sIPV (0.5ml); group 3 receives DTaP (0.5ml); group 4 receives MMR (0.5ml).

Blood samples will be collected before vaccination and 30 days after this booster immunization. Neutralization antibody will be detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of both immunization schedule will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have participated the clinical trial titled "Clinic Trial to Evaluate the Safety and Immunogenicity of Combined Immunization of sIPV and DTaP" (NCT04054882) in 2019, and have finished 3 doses of combined immunization of sIPV and DTaP;
* Subjects aged 18 months old at the date of recruitment;
* With informed consent form (ICF) signed by parent(s) or guardian(s);
* Parent(s) or guardian(s) are able to attend all planned clinical appointments and obey/follow all study instructions;
* Subjects have been vaccinated with a first dose of MMR, but have not been vaccinated with the 2nd dose of MMR and the booster (4th) dose of sIPV and DTaP;
* No less than 14 days since the last dose of vaccination;
* Axillary temperature ≤37.0℃.

Exclusion Criteria:

* With a medical history with hypersensitiveness, eclampsia, epilepsy, cerebropathia and neurological illness;
* Allergic to any ingredient of vaccine or with allergy history to any vaccine;
* Subjects with immunodeficency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(Taking orally injecting of steroid hormone);
* Administration of immunoglobulins within 30 days prior to this study;
* Acute febrile disease(temperature ≥ 37.0°C) or infectious disease;
* With a clearly diagnosed history of thrombocytopenia or other coagulopathy, may cause contraindications for subcutaneous injection;
* With any serious chronic illness, acute infectious diseases, or respiratory diseases;
* With severe cardiovascular disease, liver and kidney diseases or diabetes mellitus with complications;
* With any kind of infectious, purulent, or allergic skin diseases;
* With any other factor that makes the investigator determines the subject is unsuitable for this study.

Ages: 18 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate (sIPV) | Baseline (before vaccination) results
  determine the rate of positive seroconversion against poliovirus type I, II and III of the subjectsdetermine the rate of positive seroconversion against poliovirus type I, II and III of the subjects
Seroconversion rate (sIPV) | Results obtained 30 days after vaccination
  determine the rate of positive seroconversion against poliovirus type I, II and III of the subjectsdetermine the rate of positive seroconversion against poliovirus type I, II and III of the subjects
Seroconversion rate (DTaP) | Baseline (before vaccination) results
  determine the positive seroconversion rate of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody of the subjects
Seroconversion rate (DTaP) | Results obtained 30 days after vaccination
  determine the positive seroconversion rate of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody of the subjects
Seroconversion rate (MMR) | Baseline (before vaccination) results
  determine the positive seroconversion rate of measles, mumps, rubella antibodies of the subjects
Seroconversion rate (MMR) | Results obtained 30 days after vaccination
  determine the positive seroconversion rate of measles, mumps, rubella antibodies of the subjects
Geometric Mean Concentration (GMC) (sIPV) | Baseline (before vaccination) results
  GMCs of poliovirus type I, II and III of the subjects
Geometric Mean Concentration (GMC) (sIPV) | Results obtained 30 days after vaccination
  GMCs of poliovirus type I, II and III of the subjects
Geometric Mean Concentration (GMC) (DTaP) | Baseline (before vaccination) results
  GMCs of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody of the subjects
Geometric Mean Concentration (GMC) (DTaP) | Results obtained 30 days after vaccination
  GMCs of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody of the subjects
Geometric Mean Concentration (GMC) (MMR) | Baseline (before vaccination) results
  GMCs of measles, mumps, rubella antibodies of the subjects
Geometric Mean Concentration (GMC) (MMR) | Results obtained 30 days after vaccination
  GMCs of measles, mumps, rubella antibodies of the subjects

SECONDARY OUTCOMES:
Adverse Events Following Immunization (AEFI) | 0-6 months
  analyse the incidence of adverse events following immunization, both solicited and unsolicited

CONTACTS AND LOCATIONS:
Overall Officials: Fenyang Tang, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (3):
- China (3):
  - Anhui Provincial Center for Disease Control and Prevention, Hefei, Anhui
  - Jiangsu Province Centers for Disease Control and Prevention, Nanjing, Jiangsu
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No